CLINICAL TRIAL: NCT00433108
Title: A Double-Blind, Parallel, Randomized Comparison of Two Doses of MitoQ and Placebo for the Treatment of Patients With Raised Liver Enzymes Due to Hepatitis C
Brief Title: Trial of MitoQ for Raised Liver Enzymes Due to Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antipodean Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MTQ-HC-001
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; antioxidant; liver enzymes; ALT
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mitoquinone mesylate (MitoQ)

SUMMARY:
A Phase 2, randomized, double-blind, parallel design trial of two doses of mitoquinone mesylate (MitoQ) and of placebo in patients with chronic Hepatitis C.

MitoQ is a mitochondria-targeted antioxidant that rapidly permeates the lipid bilayer and accumulates within mitochondria in organs such as liver, brain, heart, skeletal muscle. There is strong evidence for increased oxidative stress and mitochondrial damage leading to apoptosis via caspase activation. Several studies have shown that MitoQ protects cells from apoptosis by acting as a caspase inhibitor and may be effective in reducing cell damage in liver disease.

It is hypothesised that administration of MitoQ will lower raised ALT seen in patients with chronic Hepatitis C compared with placebo. Approximately 36 patients who have been unresponsive or not suitable for interferon-based therapy will be enrolled at one centre. Treatment duration will be 28 days with 28 days post-treatment follow-up.

DETAILED DESCRIPTION:
Hepatitis C is a viral liver infection that contributes significantly to the burden of chronic liver disease. It is currently estimated that over 170 million individuals (3% of the world's population)are infected. In New Zealand, an estimated 25,000 people are living with hepatitis C virus (HCV) infection and prevalence is predicted to increase by 50% over the next 10 years. HCV is primarily spread by blood-to-blood contact. The single most important risk factor for acquiring HCV is the use of injected recreational drugs, accounting for approximately 80% of infections.

Unlike hepatitis B, no hepatitis C vaccine is currently available. In the absence of an effective vaccine the current treatment of choice is interferon and ribavirin. However, treatment of chronic HCV infection with interferon-alpha monotherapy does not achieve sustained virologic response. Therefore, it is important to develop alternative treatment strategies for patients who are unresponsive or intolerant to current antiviral therapy.

The aim of this protocol is to compare two doses of a mitochondrial antioxidant treatment (MitoQ) and placebo for the treatment of patients with raised liver enzymes due to HCV infection. Approximately 36 eligible patients with chronic HCV infection will be randomised to receive one of two doses of MitoQ or placebo in a 1:1:1 ratio. Treatment duration will be 28 days with 28 days post-treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to adhere to study requirements as evidenced by providing written informed consent before initiation of any study-related procedures
2. Aged between 18-65 years
3. Documented history of chronic HCV infection (for at least 6 months prior to study entry) as diagnosed by either:

   1. Anti-HCV positive or
   2. HCV RNA viral load positive by PCR
4. Be a non-responder to or unsuitable for interferon based therapy.
5. Have liver inflammation, as defined by either AST and/or ALT levels 2-10 x ULN on at least 1 previous occasion within the past 6 months and at Pre-treatment visit
6. alpha-fetoprotein (AFP) less than/equal to 50µg/L
7. Hemoglobin ≥100g/L, platelet count ≥75x109/L, and white blood cell count ≥1.5x109/L
8. Males, or females who are not of child-bearing potential or who are taking adequate contraceptive measures. Female patients must be postmenopausal for at least 2 years prior to the study, surgically sterile, or using effective contraception for at least 2 months prior to starting study drug and until 28 days following the last dose of study drug. Acceptable methods of birth control include hormonal contraceptives, or double-barrier methods.Negative serum pregnancy test must be documented at the Pre-treatment visit (i.e. within 14 days of starting study drug)
9. Liver biopsy within past 3 years showing stage 2 fibrosis only (i.e. excludes cirrhosis and cancer); or within past 6 years showing stage 0 or 1 (no or minimal scarring).

Exclusion Criteria:

1. Hepatocellular carcinoma (HCC) or suspicion of HCC clinically or on ultrasound (or other imaging techniques)
2. Presence of human immunodeficiency virus (HIV)
3. Co-infection with hepatitis B virus (HBV)
4. Last baseline AST and ALT level prior to Day 1 of <2.0xULN
5. Renal impairment (creatinine>1.5 x ULN) or hepatorenal syndrome
6. Chronic pancreatitis
7. Hospitalization for liver disease within 60 days of the Pre-treatment visit
8. Liver transplant recipients
9. Use of drug therapy for Hepatitis C, including the use of:

   1. drugs with presumed anti-Hepatitis C activity in the past 3 months
   2. corticosteroids in the past 30 days
   3. drugs with medium to high risk of hepatotoxicity (including alpha methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin) in the past 30 days
10. Any patient who admits to using or has a positive screening test for: amphetamines, barbiturates, pethidine, benzodiazepine, cocaine, methadone, opiates, phencyclidine or propoxyphene (unless medically prescribed and in stable doses for at least 30 days)
11. Alcohol consumption >5 units per week
12. Any patient who has received any investigational drug or device within 30 days of dosing, or who is scheduled to receive another investigational drug or device during the course of this trial
13. History of a malignancy other than treated basal cell or squamous cell carcinoma of the skin; those with a history of malignancy that has been treated with no recurrence within the last 2 years are not excluded
14. Use of antioxidants (Coenzyme Q10 and idebenone) at doses ≥300mg/day within 120 days prior to enrolment. Doses between 25-300mg/day are not an exclusion and require a 7 day washout prior to study enrolment
15. Use of dietary supplements (vitamin or mineral) at constant doses throughout the study (unless medically prescribed). Patients choosing to stop using supplements are not excluded and require a 7 day washout period prior to study enrolment
16. History of a hypersensitivity reaction to any components of the study drug or structurally similar compounds including Coenzyme Q10 and idebenone
17. Unable to swallow tablets whole.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change in serum ALT concentration at Day 28 compared with baseline

SECONDARY OUTCOMES:
Efficacy: Change in AST at Day 28 compared with baseline, change in HCV RNA viral load, plasma Mitoquinone concentration for population pharmacokinetics
Safety: Adverse events, vital signs, ECG, lab tests (biochemistry, hematology, urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Gane, MBChB, Principal Investigator — Liver Transplant Unit, Auckland City Hospital, New Zealand
Locations (2):
- New Zealand (2):
  - New Zealand Liver Unit, Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton

REFERENCES:
- [Derived] Gane EJ, Weilert F, Orr DW, Keogh GF, Gibson M, Lockhart MM, Frampton CM, Taylor KM, Smith RA, Murphy MP. The mitochondria-targeted anti-oxidant mitoquinone decreases liver damage in a phase II study of hepatitis C patients. Liver Int. 2010 Aug;30(7):1019-26. doi: 10.1111/j.1478-3231.2010.02250.x. Epub 2010 May 18. PMID 20492507